CLINICAL TRIAL: NCT03650920
Title: Pilot Investigation Using HCV Positive Liver Grafts in HCV Negative or Previously Successfully Treated Recipients
Brief Title: Hepatitis C Virus (HCV) Positive Liver Grafts in HCV Negative Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Michael Volk, Director of Transplant Hepatology, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5180105
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Liver Failure
Keywords: HCV
MeSH Terms: conditions — Liver Failure | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recipient of HCV positive liver graft (Experimental): A single center, open-label, pilot study examining 10 adult HCV negative liver transplant subjects who receive an HCV infected graft. Target start date for antiviral therapy will be within 3 months after liver transplantation, unless extenuating clinical circumstances arise (such as fibrosing cholestatic HCV, which would prompt earlier treatment, or non-hepatic comorbidities which would prompt delay in treatment).
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — A HCV negative or previously successfully treated recipient with a HCV positive liver graft

SUMMARY:
To provide proof-of-concept data on the efficacy/safety of transplanting HCV positive donor grafts in HCV sero-negative liver recipients who are currently listed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 and older
* Active on the transplant list
* Donor organ with Antibody and nucleic acid test (NAT) positive for HCV
* Graft with F2 fibrosis or less at time of explant
* HCV negative recipient; this includes patients who never had HCV and those with HCV previously eradicated with antiviral therapy. The latter is defined as those with undetectable HCV viral load at least 3 months since stopping therapy.
* Willing and able to provide written informed consent or for those subjects where hepatic encephalopathy affects their ability to provide initial or ongoing consent, has an appropriate and legally-authorized representative willing and able to provide consent on behalf of the subject

Exclusion Criteria:

* Participants co-infected with HIV
* Donor previously treated with a non-structural protein 5A (NS5a) containing regimen (if treatment history of donor known)
* Known allergies or hypersensitivity to direct acting antiviral drug (DAA) or ribavirin (RBV)
* Pregnancy and/or actively breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Patient survival rate | From the date of transplant through the last day of 15 month post transplant
  Will track all subjects post transplant for 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Volk, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Transplant Institute, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levitsky J, Formica RN, Bloom RD, Charlton M, Curry M, Friedewald J, Friedman J, Goldberg D, Hall S, Ison M, Kaiser T, Klassen D, Klintmalm G, Kobashigawa J, Liapakis A, O'Conner K, Reese P, Stewart D, Terrault N, Theodoropoulos N, Trotter J, Verna E, Volk M. The American Society of Transplantation Consensus Conference on the Use of Hepatitis C Viremic Donors in Solid Organ Transplantation. Am J Transplant. 2017 Nov;17(11):2790-2802. doi: 10.1111/ajt.14381. Epub 2017 Jul 1. PMID 28556422
- See also: Use of Hepatitis C Viremic Donors in Solid Organ Transplantation — https://www.ncbi.nlm.nih.gov/pubmed/28556422